CLINICAL TRIAL: NCT01417585
Title: A Randomized Controlled Trial of a Client-centered Intervention Aiming to Improve Functioning in Daily Life After Stroke
Brief Title: A Trial of a Client-centered Intervention Aiming to Improve Functioning in Daily Life After Stroke
Acronym: LAS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Council for Working Life and Social Research (Other); The Swedish Brain Foundation (Hjärnfonden) (Unknown); Stroke-Riksförbundet (Unknown); Region Stockholm (Other Government); Uppsala County Council, Sweden (Other Government); Uppsala-Örebro Regional Research Council (Other)
Responsible Party: Principal Investigator, Lena von Koch, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2009/727-31/1
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2012-01

CONDITIONS: Stroke; Physical Disability; Multiple Disability
Keywords: Activities of daily living; Caregiver burden; Client centered; Life satisfaction; Participation; Patient satisfaction; Rehabilitation; Self rated impact of stroke; Stroke
MeSH Terms: conditions — Stroke; Caregiver Burden; Personal Satisfaction; Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Client-centered ADL intervention — Client-centered ADL refers to rehabilitation of activities of daily living specifically guided by the needs as expressed by the client/patient and her/his significant others, a process that specifically aims to support the client by taking the client's goals and views as the guide for the rehabilitation process.
Behavioral: Usual ADL intervention — The variation of strategies and ways to conduct usual ADL rehabilitation according to the routines and praxis of the participating rehabilitation units randomized to supply the control condition.

SUMMARY:
This is a cluster randomized controlled trial in which client-centered rehabilitation of activities of daily living (CADL) will be compared to usual rehabilitation of activities of daily living (UADL) regarding participation in activities of daily living, independence in activities of daily living and life satisfaction during the first year after stroke. In addition use of health services, caregiver burden and significant others' life satisfaction will be studied. Study design, methods and power analysis are based on our previous pilot study. Participating rehabilitation centers in the counties of Stockholm, Uppsala and Gavleborg have been randomized to supply CADL or UADL. Patients are included who are: < 3 months after stroke, dependent in at least two activities of daily living, understand instructions and referred to a participating rehabilitation unit. Data are collected at baseline, 3, 6 and 12 months. For sufficient power 280 participants will be included. In addition qualitative longitudinal studies will be performed in order to describe how CADL is integrated.

ELIGIBILITY:
Inclusion Criteria:

* < 3 months after stroke
* Dependent in at least two activities of daily living
* Able to understand instructions
* Referred to a participating rehabilitation unit.

Exclusion Criteria:

* Diagnosed dementia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Perceived participation | 12 months

SECONDARY OUTCOMES:
Life satisfaction | 3 and 12 months
Utilization of health care and health related services | During one year after inclusion
Fatigue | baseline, 3, 6 and 12 months
Caregiver burden | 3 and 12 months
Self rated impact of stroke | 3, 6 and 12 months
  Stroke Impact Scale
Activities of daily living | baseline, 3, 6 and 12 months
Satisfaction with care | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Tham, PhD, Study Chair — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Tistad M, Flink M, Ytterberg C, Eriksson G, Guidetti S, Tham K, von Koch L. Resource use of healthcare services 1 year after stroke: a secondary analysis of a cluster-randomised controlled trial of a client-centred activities of daily living intervention. BMJ Open. 2018 Aug 5;8(8):e022222. doi: 10.1136/bmjopen-2018-022222. PMID 30082359